CLINICAL TRIAL: NCT06089434
Title: Transesophageal Echocardiography (TEE) and Dysphagia in Lung Transplantation (LT)
Brief Title: TEE and Dysphagia in Lung Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jacques Neelankavil, Principal Investigator and Professor of Clinical Anesthesiology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-000600
Record Dates: First submitted 2023-09-26; First posted 2023-10-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Lung Transplant; Dysphagia
Keywords: Lung Transplantation; Dysphagia; Transesophageal Echocardiography (TEE); Outcomes
MeSH Terms: conditions — Deglutition Disorders | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transesophageal Echocardiography (TEE) with limited number of TEE clips (Experimental): The intervention group would limit the number of TEE clips per case.
  Interventions: Diagnostic Test: Transesophageal Echocardiography (TEE) with limited number of TEE clips
- Transesophageal Echocardiography (TEE) with number of TEE clips per attending anesthesiologist (Other): The control group would leave the number of TEE clips to the discretion of the attending anesthesiologist.
  Interventions: Diagnostic Test: Transesophageal Echocardiography (TEE) with number of TEE clips per attending anesthesiologist

INTERVENTIONS:
Diagnostic Test: Transesophageal Echocardiography (TEE) with limited number of TEE clips — The intervention group would be limited to fewer than 20 TEE clips per case (versus the average of ~ 80-100 TEE clips per case).
  Arms: Transesophageal Echocardiography (TEE) with limited number of TEE clips
Diagnostic Test: Transesophageal Echocardiography (TEE) with number of TEE clips per attending anesthesiologist — The control group would leave the number of TEE clips to the discretion of the attending anesthesiologist.
  Arms: Transesophageal Echocardiography (TEE) with number of TEE clips per attending anesthesiologist

SUMMARY:
The primary outcome of this study is dysphagia (difficulty swallowing) on postoperative speech and swallow evaluation following lung transplantation.

Transesophageal echocardiography (TEE) (creates pictures of the heart from inside the participants body) is routinely performed for all lung transplantations at the University of California, Los Angeles (UCLA) and it is the standard of care. Patients are randomized to two groups. The intervention group would limit the number of TEE clips (# pictures taken) per case. The control group would leave the number of TEE clips to the discretion of the attending anesthesiologist.

The investigators hypothesize that reduction in TEE imaging during lung transplantation will reduce dysphagia.

DETAILED DESCRIPTION:
Dysphagia is a common complication after cardiac surgery and specifically after lung transplantation. The incidence of dysphagia after lung transplantation is approximately 40-50%. Dysphagia after cardiac surgery leads to a significant increase in mortality, morbidity, cost, and length of stay. There are several risk factors that have been identified retrospectively including patient comorbidities, length of surgery, length of intubation, and number of TEE clips obtained during surgery. Many of these risk factors are not modifiable, however, the number of TEE clips obtained is a potential area for intervention. Retrospective studies demonstrate that a high number of TEE clips may be associated with dysphagia postoperatively. TEE should not be completely eliminated from these procedures because it adds value for patient management and the diagnosis of intraoperative complications.

This is a prospective, cluster randomized study for adult patients undergoing single and double lung transplantation. Groups will be randomized by month. The primary outcome of the study is dysphagia on postoperative speech and swallow evaluation.

TEE is routinely performed for all lung transplantation at UCLA and it is the standard of care. Patients would be randomized to two groups. The intervention group would be limited to fewer than 20 TEE clips per case. The control group would leave the number of TEE clips to the discretion of the attending anesthesiologist (average ~80-100 TEE clips per case). The current standard of care is to leave the number of TEE clips to the discretion of the attending anesthesiologist (the control arm). The attending anesthesiologist has the ability to obtain more TEE clips in the intervention arm if they feel it will be beneficial to patient care.

The postoperative speech and swallow evaluation is standard of care for all lung transplant recipients and would be done regardless of participation in the study. This is a bedside evaluation done by a speech/language therapist after the patient has been extubated, usually performed on postoperative day (POD) 1.

Data will also be collected and recorded from the medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Single or double lung transplantation

Exclusion Criteria:

1. Contraindications to TEE including:

   * perforated esophagus;
   * esophageal stricture;
   * esophageal tumor; and
   * history of an esophagectomy
2. Patients that require a tracheostomy postoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dysphagia | Postoperative Day 1 (POD1)
  Dysphagia on the postoperative speech and swallow evaluation. Dysphagia is classified into 3 major classifications: swallowing without limitations, swallowing with limitations, and inability to swallow.

SECONDARY OUTCOMES:
Mortality | POD0 until discharge from the hospital. An average of 5-10 days until discharge from the hospital. A maximum of 30 days for in-hospital mortality.
  In-hospital mortality
Length of Intubation | From time of intubation until time to extubation, in hours, on average POD0 or POD1.
  Number of hours intubated from POD0 to extubation.
Length of intensive care unit (ICU) Stay | From time of admission to the ICU (POD0) until discharge from the ICU. An average of 3-5 days.
  Number of days in the ICU from POD0 to discharge from the ICU.
Length of Hospital Stay | From time of admission to the ICU (POD0) until discharge from the hospital, An average of 5-10 days.
  Number of days in the hospital from POD0 to discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: J.Prince Neelankavil, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology & Perioperative Medicine, Los Angeles, California, United States